CLINICAL TRIAL: NCT06344689
Title: The Surgical Correction of Cicatricial Ectropion: a Retrospective Study
Brief Title: Surgical Correction of Cicatricial Ectropion
Status: Completed | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Lin Lu, PhD., Doctor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: SH9H-2023-T477
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Patients With Cicatricial Ectropion; Over 18-year-old; With Complete Clinical Record
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ectropion underwent surgical treatment.
  Interventions: Other: Surgical treatment

INTERVENTIONS:
Other: Surgical treatment — Patients underwent surgical treatment of ectropion were included in this study.

SUMMARY:
The main purpose of this study is to verify and compare the treatment effects of scarred ectropion surgery, perform statistical descriptions, compare patients undergoing tarsal strip and skin flap procedures with those undergoing simple skin flap treatment, and compare their pre- and post-operative Ectropion Grading Scale (EGS) and subjective and objective symptom changes.

Secondary Objective: To observe the incidence and resolution of complications after lower eyelid ectropion surgery. Compare postoperative effects among patients of different ages undergoing the same surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients with Cicatricial Ectropion;
* over 18-year-old;
* with complete clinical record.

Exclusion Criteria:

* patients with severe complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ectropion underwent surgical treatment in our center.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Ectropion Grading Scale | preoperative and one-year posttreatment
  The EGS describes the severity of the ectropion, with higher score for more severe ectropion.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai ninth people's hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided